CLINICAL TRIAL: NCT07022899
Title: Laser and Phenol Treatment for Pilonidal Sinus: Outcomes of Monotherapy and Combined Approach
Brief Title: Laser and Phenol Treatment for Pilonidal Sinus
Status: Active, not recruiting | Type: Observational
Sponsor: Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adnan Gundogdu, MD, Sehit Prof. Dr. Ilhan Varank Sancaktepe Training and Research Hospital
Other Study IDs: Ivstrh_pilonidal
Record Dates: First submitted 2025-06-08; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Pilonidal Sinus Treatment
Keywords: Pilonidal Cyst Pilonidal Abscess Sacrococcygeal Pilonidal Sinus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Laser Therapy Group Group Type: Other: Patients receiving diode laser treatment alone for pilonidal sinus disease
- Phenol Treatment Group: Patients receiving crystallized phenol application alone for pilonidal sinus disease
- Combined Treatment Group: Patients receiving both laser therapy and phenol treatment in combination for pilonidal sinus disease

SUMMARY:
This study compares three different treatments for pilonidal sinus disease to determine which approach provides the best outcomes for patients.

Pilonidal sinus is a condition where a small hole or tunnel forms in the skin at the top of the buttocks. It happens when hair gets trapped under the skin, causing pain, swelling, and infection. This condition mainly affects young adults and can interfere with work and daily activities.

The study compares three minimally invasive treatments:

1. Laser therapy alone: A thin laser fiber is inserted into the sinus to destroy the lining and close the tunnel using local anesthesia as an outpatient procedure.
2. Phenol treatment alone: A chemical solution (phenol) is injected into the sinus to make it close and heal, done with local anesthesia in the clinic.
3. Combined laser and phenol therapy: Both treatments are used together for potentially better healing with lower recurrence rates.

Researchers will measure healing rates, healing time, recurrence rates, pain levels, complications, patient satisfaction, and return to normal activities.

This research is important because there is no single "best" treatment for pilonidal sinus. Traditional surgery often requires general anesthesia, hospital stays, large wounds taking months to heal, significant scarring, long work absence, and high recurrence rates up to 30%.

These newer treatments offer faster healing, less pain and scarring, quicker return to normal life, and lower recurrence chance. By comparing these approaches directly, this study will help doctors and patients make better treatment decisions based on scientific evidence.

This is a prospective observational cohort study following patients who receive one of these three treatments. The study will include adults with pilonidal sinus disease suitable for minimally invasive treatment.

DETAILED DESCRIPTION:
Detailed Description şu şekilde olmalı (sample size dahil):

STUDY DESIGN AND METHODOLOGY

This prospective observational cohort study will be conducted at Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, Department of General Surgery. The study aims to compare the clinical outcomes of three different minimally invasive treatment approaches for pilonidal sinus disease.

TREATMENT GROUPS

Group 1 - Laser Therapy: Patients will receive diode laser treatment using a radial fiber inserted into the pilonidal sinus tract. The procedure is performed under local anesthesia with lidocaine injection.

Group 2 - Phenol Treatment: Patients will receive crystallized phenol application into the sinus cavity after debridement of hair and debris. The procedure is performed under local anesthesia.

Group 3 - Combined Treatment: Patients will receive both laser therapy followed by phenol application in the same session under local anesthesia.

SAMPLE SIZE

This is a pilot comparative study designed to evaluate the feasibility and preliminary efficacy of three treatment approaches. Sample size will be determined based on patient availability and recruitment capacity during the study period. All eligible patients meeting inclusion criteria will be enrolled consecutively.

FOLLOW-UP SCHEDULE

Patients will be evaluated at 1 week, 1 month, 3 months, 6 months, and 12 months post-treatment.

PRIMARY ENDPOINTS

* Complete healing rate (absence of discharge, pain, and complete epithelialization)
* Recurrence rate at 12 months

SECONDARY ENDPOINTS

* Time to complete healing
* Post-operative pain scores (VAS)
* Complication rates
* Patient satisfaction scores
* Return to normal activities
* Quality of life assessment

STATISTICAL ANALYSIS

Categorical variables will be analyzed using Chi-square test. Continuous variables will be analyzed using appropriate parametric or non-parametric tests. Kaplan-Meier survival analysis will be used for time-to-healing assessment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Diagnosed chronic pilonidal sinus disease confirmed by clinical examination
* Suitable for minimally invasive treatment approaches
* Ability to provide informed consent
* Willingness to comply with follow-up schedule
* No contraindications to local anesthesia

Exclusion Criteria:

* Active acute pilonidal abscess requiring emergency drainage
* Previous pilonidal sinus surgery or treatment
* Pregnancy or breastfeeding
* Immunocompromised patients (diabetes mellitus, immunosuppressive therapy, chronic corticosteroid use)
* Malignancy in the sacrococcygeal region
* Bleeding disorders or anticoagulant therapy that cannot be discontinued
* Allergy to local anesthetics (lidocaine)
* Mental incapacity or psychiatric illness preventing informed consent
* Geographic inaccessibility for follow-up visits

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with chronic pilonidal sinus disease seeking treatment at Sancaktepe Şehit Prof. Dr. İlhan Varank Training and Research Hospital, Department of General Surgery.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2026-06-25 (Estimated)

PRIMARY OUTCOMES:
Complete Healing Rate | 6 months
  Complete Healing Rate
Recurrence Rate | 12 months
  Percentage of patients experiencing recurrence of pilonidal sinus disease defined as reappearance of symptoms, discharge, or new sinus formation at the treatment site

SECONDARY OUTCOMES:
Time to Complete Healing | Up to 12 months
  Time in weeks from treatment to complete healing
Post-operative Pain Score | 1 week, 1 month, 3 months
  Pain intensity measured using Visual Analog Scale (VAS) ranging from 0-10
Complication Rate | 12 months
  Percentage of patients experiencing treatment-related complications

CONTACTS AND LOCATIONS:
Locations (1):
- Sancaktepe Sehit Prof. Dr. Ilhan Varank Training and Research Hospital, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared due to patient privacy protection requirements under Turkish data protection laws and the small sample size of this single-center study. Study results will be shared through scientific publications.